CLINICAL TRIAL: NCT05471297
Title: Effects of Physical, Psychosocial and Dual-career Loads on Injuries and Illnesses Among Elite Handball Players
Brief Title: Loads, Injuries and Illnesses Among Elite Handball Players
Acronym: PPDC-2022
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Armin Paravlic, Supervisor, University of Ljubljana
Other Study IDs: PPDC-2022
Record Dates: First submitted 2022-07-17; First posted 2022-07-22 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Injuries; Illnesses Systemic; Illness, Chronic; Illnesses, Occupational; Psychological; Physical Illness; Physical Stress; Physical Injury; Physical Trauma; Social Stress; Athletic Injuries
MeSH Terms: conditions — Wounds and Injuries; Chronic Disease; Occupational Diseases; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken to investigate the levels of testosterone, cortisol and IgA hormones during a single competitive season
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Handball players: Professional handball players
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no any intervention

SUMMARY:
Primary goal of the research is to determine whether injury/illness occurrence is influenced by the academic, training and competition loads, as well as the overall load (sum of academic/work, training and competition loads) in elite handball athletes To examine whether subjective measures of perceived overall stress correlate with objectively measured levels of stress.

Determine the benefits of certain biomarkers to monitor stress, load and injury/illness occurrence in athletes.

DETAILED DESCRIPTION:
The current structure and organizational initiatives do not meet the needs of athletes as they face different challenges throughout their careers. There is a need for better health surveillance, load monitoring and support services with a focus on injury/illnesses prevention and rehabilitation. The main goal of the research is to determine how specific loads affect the occurrence of injuries and illnesses in elite handball players and how much of the total load an athlete can withstand before an injury/illness occurs. Thus, the study will attempt to identify athletes at risk of injury/illness by monitoring their workload with subjective (perceived stress) and objective (biomarkers, hours of workload) measurements. One of the goals is also to determine the correlation between objective measures of stress (biomarkers) and subjective measures of stress (athlete's stress assessment). The results will not only be important for the medical and sports community for development of new injury prevention and rehabilitation strategies, but also for structuring the correct policy recommendations for athletes' general health. The research will be carried out on approx. 250 elite handball players (the entire 1st men's handball league) during one handball season. In addition to other parameters (monitoring of load, injuries and illnesses), blood samples will be taken from athletes at five time points according to their training cycle.

ELIGIBILITY:
Inclusion Criteria:

* At least national-level handball players above 18 years of age, who are in a dual-career setting.
* Handball players older than 18 years old, who are competing at least at national level and are not in a dual-career setting will be matched by their demographic characteristics and included in the control group.

Exclusion Criteria:

* Not fulfilling inclusion critieria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first league handball players
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The Oslo Sports Trauma Research Center Questionnaire on Health Problems (OSTRC) | 12 months
  Injury and illness questionnaire
Load | 12 months
  PHYSICAL, PSYCHOSOCIAL AND DUAL-CAREER loads

SECONDARY OUTCOMES:
Biomarkers | 12 months
  testosterone, cortisol, Immunoglobulin A (IgA)
Life Events Survey for Collegiate Athletes (LESCA) questionnaire | 12 months
  Life Events Survey for Collegiate Athletes questionnaire

OTHER OUTCOMES:
Body composition | 12 months
  Body composition measurements with bio-impedance

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Drole, MSc, Principal Investigator — Faculty of Sport, University of Ljubljana
Locations (2):
- Slovenia (2):
  - Faculty of Sport, Ljubljana, Slovenia
  - Handball Clubs, Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon the reasonable request to principal investigator

REFERENCES:
- [Background] Drole K, Paravlic A, Steffen K, Doupona M. Effects of physical, psychosocial and dual-career loads on injuries and illnesses among elite handball players: protocol of prospective cohort study. BMJ Open. 2023 Mar 2;13(3):e069104. doi: 10.1136/bmjopen-2022-069104. PMID 36863744
- [Derived] Drole K, Busch A, Paravlic A, Doupona M, Steffen K. Prevalence, incidence and burden of health problems across playing positions in elite male handball players: a 45-week prospective cohort study. BMJ Open Sport Exerc Med. 2025 Apr 5;11(2):e002460. doi: 10.1136/bmjsem-2025-002460. eCollection 2025. PMID 40195973
- [Derived] Drole K, Steffen K, Paravlic A. Slovenian Translation, Cross-Cultural Adaptation, and Content Validation of the Updated Oslo Sports Trauma Research Center Questionnaire on Health Problems (OSTRC-H2). Orthop J Sports Med. 2024 Nov 13;12(11):23259671241287767. doi: 10.1177/23259671241287767. eCollection 2024 Nov. PMID 39539687
- See also: Link to a study protocol — https://bmjopen.bmj.com/content/13/3/e069104